CLINICAL TRIAL: NCT00338182
Title: A Phase I, Open-Label, Multi-Centre Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD1152 Given as a 2-hour or 48-hour Intravenous Infusions in Patients With Advanced Solid Malignancies
Brief Title: AZD1152 in Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1531C00002
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Tumors
Keywords: Solid tumor
MeSH Terms: conditions — Neoplasms

ARMS (1):
- AZD1152 (Experimental): AZD1152 treatment given for 2 days every 14 days (2 treatment days followed by 12 days off treatment)
  Interventions: Drug: AZD1152 part A; Drug: AZD1152 part B

INTERVENTIONS:
Drug: AZD1152 part A — 48-hour continuous intravenous infusion
Drug: AZD1152 part B — 2-hour intravenous infusion

SUMMARY:
The primary purpose of this protocol is to investigate the safety and tolerability of AZD1152 when given as a continuous 48-hour infusion every 14 days and as a 2-hour infusion for 2 consecutive days every 14 days in patients with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of a solid, malignant tumour
* At least one measurable or non-measurable site of disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

Exclusion Criteria:

* Participation in an investigational drug study within the 21 days prior to therapy or those who have not recovered from the effects of an investigational study drug
* Recent major surgery within 4 weeks prior to entry into the study

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-05-23 (Actual); Primary Completion 2008-06-06 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events (including adverse events detected via laboratory assessment, vital signs and ECG) | Throughout the study. Approximately 9 months for most patients.
  Safety and tolerability will be assessed through the incidence of adverse events. Adverse events will include significant findings on vital signs, clinical chemistry/haematology, coagulation parameters and electrocardiograms (ECGs).

SECONDARY OUTCOMES:
Assessment of pharmacodynamic biomarker changes | Biopsies of tumour at baseline and Cycle 1 [at pre-dose, after Screening to Day 1; and between Days 16-19 (preferrably within 24 hours of completing infusions on Day 17 (Part A) and Day 16 (Part B).]
  Evaluation of AZD1152 activity in the tumour by assessment of pharmacodynamic biomarker changes which may include, but are not limited to biomarkers of Aurora kinase activity.

CONTACTS AND LOCATIONS:
Overall Officials: Emerging Oncology Medical Science Director, MD, Study Director — AstraZeneca
Locations (2):
- United States (2):
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1163&filename=CSR-D1531C00002.pdf
- See also: CSR-D1531C00002.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1163&filename=CSR-D1531C00002.pdf